CLINICAL TRIAL: NCT06458881
Title: EFFICACY OF A MIXTURE OF SIMETHICONE AND TYNDALLIZED BACILLUS COAGULANS IN INFANT COLIC: A PILOT STUDY
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Marina Russo, Dott. Marina Russo, Federico II University
Other Study IDs: 196/2023
Record Dates: First submitted 2024-06-11; First posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Infant Colic
MeSH Terms: conditions — Colic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Combination Product: Mixture of Simethicone and Tyndallized Bacillus Coagulans — . Enrolled infants were treated for 28 days with a mixture of Tyndallized B. Coagulans and Simethicone: 20 drops, four times a day. At enrolment, clinical and dietary history, obstetrical data and anthropometry were recorded. The subjects were classified as having IC based on their parents' responses to the validated questionnaires regarding IC according to Rome IV criteria.

SUMMARY:
: A pilot study was conducted on a group of 41 infants with diagnosis of Infant Colic according to Rome IV criteria. We administered to all the enrolled infants a mixture of Tyndallized bacillus coagulans and Simethicone for 28 days. The primary outcome was the mean infant crying duration at 28th day. The secondary outcome was the improvement in the quality of sleep and infants' and parents' quality of life

DETAILED DESCRIPTION:
This pilot study is a prospective study coordinated by the Department of Translational Medicine, Section of Pediatrics, University of Naples "Federico II", whereas infants were recruited by 8 general pediatricians belonging to the Pediatrics Investigator Committee of Campania Region, Italy. Inclusion criteria were: full term infants (>_37 weeks gestation at birth; 5-min Apgar score >_7; Birth weight >_2500 g), aged <12 months, diagnosed with IC according to Rome IV criteria [1], breast- and formulafed infants. The parents of the infants participating in the study were supplied with the mixture of Tyndallized B. Coagulans and Simethicone. The Institutional Review Board of Campania 3 approved the research protocol. All parents gave written informed consent. Enrolled infants were treated for 28 days with a mixture of Tyndallized B. Coagulans and Simethicone: 20 drops, four times a day. At enrolment, clinical and dietary history, obstetrical data and anthropometry were recorded. The subjects were classified as having IC based on their parents' responses to the validated questionnaires regarding IC according to Rome IV criteria. The parents were also asked to fill in the following questionnaires: 1) Baby's Day Diary on daily crying and infant sleep duration [21]; 2) a scale (visual analogue scale, VAS, 0e10) for parents' quality of life, a questionnaire on infant's quality of life; 3) a form for stool frequency and consistency; 4) a scale for parental perception of colic severity (VAS 0e10) and 5) a scale for parental perception of sleep quality (VAS 0 e10). Infants were evaluated by a physician for follow-up visits at week 4. During the visits, physical examination was performed and information regarding drugs administration, number and site of infections and eventual adverse medical events were recorded. Moreover, parents had to fill: 3) the questionnaire on infant's quality of life; 4) a review of stool frequency and consistency; 5) the parental perception of colic severity (VAS 0e10) and 6) the parental perception of sleep quality (VAS 0e10). All the authors had access to the study data. Compliance was assessed by evaluating the diary provided by the parents.

Outcomes The primary endpoint was the infant crying duration at 28 days. Treatment success was defined as at least 50% reduction in crying time from baseline to day 28 postintervention. Secondary endpoints included: infant sleep duration at 28 days post-intervention, mean scores on a standardized measure of parents' and infants' quality of life, changes in stool consistency, number of episodes of infant colic per day, parental perception of colic severity (VAS 0-10), parental perception of quality of life (VAS0-10).

ELIGIBILITY:
Inclusion Criteria:

- Inclusion criteria were: full term infants (>_37 weeks gestation at birth; 5-min Apgar score >_7; Birth weight >_2500 g), aged <12 months, diagnosed with IC according to Rome IV criteria [1], breast- and formulafed infants.

Exclusion Criteria:

-

Ages: 1 Month to 12 Months | Sex: All
Age Groups: Child
Gender Based: Yes
Study Population: Sample size determination was guided by the primary objective of the study and was based on the approach described in Sung et al. (12), using data subsequently published in Sung et al. (13). Specifically, we considered as a comparison base, and as a proxy for a physiological reduction in crying, the success rate (defined as a reduction in crying time by at least 50%) in the placebo group, which Sung et al. (13) reported to be 39%. In comparison, the success rate observed in subjects treated with probiotics was 66%. Therefore, a sample size of 37 subjects was found sufficient to achieve 90% power to detect a success rate of 0.66 (assuming under the null hypothesis a proportion of 0.39), using a two-sided exact test with a 5% significance level. Considering a dropout rate of 10%, 41 patients were enrolled.
Sampling Method: Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
The primary endpoint was the infant crying duration at 28 days. | reatment success was defined as at least 50% reduction in crying time from baseline to day 28 postintervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Marina Russo, Napoli, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Saviano M, Russo M, Buono P, La Pietra M, Sorrentino E, Chianese A, Ementato S, Illiano G, Napolitano G, Dolce P, Staiano A. Efficacy of a mixture of simethicone and tyndallized bacillus coagulans in infant colic: a pilot study on behalf of Italian Society of Pediatrics (SIP). Ital J Pediatr. 2025 Nov 12;51(1):300. doi: 10.1186/s13052-025-02140-2. PMID 41225617